CLINICAL TRIAL: NCT04270786
Title: Phase III Randomized Study of Early De-escalation of Empirical Antibiotics Treatment for Neutropenic Fever in Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Early De-escalation of Empirical Antibiotics Treatment for Neutropenic Fever
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood and Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-BMT-Antibio
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Safety Issues
Keywords: neutropenic fever, empiric, antibiotics
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early de-escalation (Experimental): In the experiment arm, empirical antibiotics will be stopped and levofloxacin prophylaxis will be resumed in case of afebrile after 72 hours.
  Interventions: Procedure: Early de-escalation
- Standard (Other): In the control group, empirical antibiotics will be continue until recovery of neutropenia or at least 7 days as standard clinical practice.
  Interventions: Procedure: Standard

INTERVENTIONS:
Procedure: Early de-escalation — In de-escalating group, the empirical antibiotics will be stopped and then prophylaxis levofloxacin will be resumed.
  Arms: Early de-escalation
Procedure: Standard — In the control arm, empirical antibiotics will be continue until recpvery of neutropenia or at least 7 days after afebrile.
  Arms: Standard

SUMMARY:
This is a randomized study to evaluate the safety and feasibility of early de-escalation of empirical antibiotics treatment in neutropenic fever patients undergoing hematopoietic stem cell transplantation (HSCT). In case of afebrile for 72 hours with empirical antibiotics treatment, patients will be randomized into 2 groups. In the early de-escalation group, antibiotics treatment will be stopped and prophylaxis with levofloxacin will be resumed. In the control group, the empirical treatment will continue until recovery of neutropenia or at least for 7 days.

DETAILED DESCRIPTION:
This is a randomized study to evaluate the safety and feasibility of early de-escalation treatment of empyrical antibiotics treatment in neutropenic fever patients undergoing hematopoietic stem cell transplantation (HSCT). All patients undergoing HSCT will receive levofloxacin as regular prophylaxis. After patients develop neutropenia fever, the empirical antibiotics protocol will be impenem. In case of persistent for 48 hours, vancomycin will be added. If afebrile is achieved for 72 hours, all patients will randomized into early de-escalating group or control group. In de-escalating group, the empirical antibiotics treatment will be stopped and then levofloxacin prophylaxis will be resumed. In the control group, the empirical antibiotics treatment will be continue until recovery of neutropenia or at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18，patients undergo hematopoietic stem cells
* Patients with neutropenic fever: T≥38.5°C once or T≥38°C twice a day with ANC <0.5x109/L or predicted to be <0.5x109/L in 24 ~48 hours；
* Patients achieved afebrile （T<37.5°C）for at least 72 hours；
* Inform consent given

Exclusion Criteria:

* Patients with neutropenic fever with documented blood stream infection, skin and soft tissue infection, pneumonia and catheter associated infection.
* Patients with septic shock
* Levofloaxin allergy or contra-indication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Days of no empirical antibiotics treatment | 28 days
  days from start of empirical antibiotics to end of study minus days with empirical antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Jiong hu, Principal Investigator — Ruijin Hospital
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, Shanghai Municipality, China